CLINICAL TRIAL: NCT02416622
Title: A Multiple-Site, Phase 1/2, Safety and Efficacy Trial of a Recombinant Adeno-associated Virus Vector Expressing Retinoschisin (rAAV2tYF-CB-hRS1) in Patients With X-linked Retinoschisis
Brief Title: Safety and Efficacy of rAAV-hRS1 in Patients With X-linked Retinoschisis (XLRS)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beacon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGTC-RS1-001
Record Dates: First submitted 2015-04-02; First posted 2015-04-15 (Estimated); Results first posted 2020-07-01 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: X-linked Retinoschisis
Keywords: XLRS; maculoschisis; retinal degeneration; RS1; adeno-associated virus; gene therapy; AAV
MeSH Terms: conditions — Retinoschisis; Retinal Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Groups 1A and 1B (Experimental): Subjects at least 18 y/o treated with a lower dose of rAAV2tYF-CB-hRS1 study drug.
  Interventions: Biological: rAAV2tYF-CB-hRS1
- Groups 2 and 2A (Experimental): Subjects at least 6 y/o treated with a middle dose of rAAV2tYF-CB-hRS1 study drug.
  Interventions: Biological: rAAV2tYF-CB-hRS1
- Group 3 (Experimental): Subjects at least 18 y/o treated with a higher dose of rAAV2tYF-CB-hRS1 study drug.
  Interventions: Biological: rAAV2tYF-CB-hRS1
- Group 4 (Experimental): Subjects at least 6 y/o treated with a maximum tolerated dose of rAAV2tYF-CB-hRS1 study drug determined for Groups 1A, 1B, 2 and 3.
  Interventions: Biological: rAAV2tYF-CB-hRS1

INTERVENTIONS:
Biological: rAAV2tYF-CB-hRS1 — adeno-associated virus vector expressing retinoschisin

SUMMARY:
This study will evaluate the safety and efficacy of a recombinant adeno-associated virus vector expressing retinoschisin (rAAV2tYF-CB-hRS1) in patients with X-linked retinoschisis. Up to 27 participants will be enrolled and 3 dose levels will be evaluated in a dose escalation format.

DETAILED DESCRIPTION:
This will be a non-randomized, open label, Phase 1/2 dose escalation study.

Up to 27 participants will be enrolled. Each participant will receive the study agent by intravitreal injection in one eye on a single occasion. Enrollment will begin with the lowest dose and will proceed to higher doses only after review of safety data by a Data and Safety Monitoring Committee (DSMC). Participants in the dose escalation phase will be ≥ 18 years of age. After the maximum tolerated dose is identified individuals ≥ 6 years of age will be enrolled.

Safety will be measured by the number and proportion of participants experiencing adverse events and immune response to RS1. Efficacy will be measured by evaluation of changes in visual function and schisis cavity size.

ELIGIBILITY:
Inclusion Criteria include:

1. Retinal disease consistent with a diagnosis of XLRS and documented mutations in the RS1 gene
2. Male individual at least 18 years of age (dose escalation phase) or at least 6 years of age (maximum tolerated dose phase),
3. Able to perform tests of visual and retinal function,
4. Visual acuity specified for each group
5. Not treated with CAIs currently or within 3 months prior to study enrollment,
6. Have acceptable laboratory parameters.

Exclusion Criteria include:

1. Prior receipt of any AAV gene therapy product,
2. Pre-existing eye conditions that would preclude the planned intravitreal injection or interfere with interpretation of study endpoints or complications of vector administration.

Min Age: 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2023-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Heah, MD, Study Director — Applied Genetics Technologies Corporation
Locations (9):
- United States (9):
  - University of California San Francisco, Dept. of Ophthalmology, San Francisco, California
  - University of Miami - Miller School of Medicine Bascom Palmer Eye Institute, Miami, Florida
  - The Wilmer Eye Institute, Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - University of Michigan Kellogg Eye Center, Ann Arbor, Michigan
  - Duke Eye Center, Duke University Medical Center, Durham, North Carolina
  - Casey Eye Institute, Oregon Health and Sciences University, Portland, Oregon
  - Retina Foundation of the Southwest, Dallas, Texas
  - Baylor College of Medicine, Alkek Eye Center, Houston, Texas

REFERENCES:
- [Background] Molday RS, Kellner U, Weber BH. X-linked juvenile retinoschisis: clinical diagnosis, genetic analysis, and molecular mechanisms. Prog Retin Eye Res. 2012 May;31(3):195-212. doi: 10.1016/j.preteyeres.2011.12.002. Epub 2012 Jan 3. PMID 22245536
- See also: AGTC website — http://agtc.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No participants have completed the study at this time because the study is ongoing (overall status: active, not recruiting). All enrolled participants are in long term follow-up.
Groups:
- rAAV2tYF-CB-hRS1 1 x 10^11 vg Per Eye: Group 1A/1B: Adult participants were administered a single intravitreal (IVT) injection of rAAV2tYF-CB-hRS1, once in the study eye, at a dose of 1 x 10^11 vg/eye and followed for a minimum of 12 months after dose administration.
- rAAV2tYF-CB-hRS1 3 x 10^11 vg Per Eye: Group 2/2A: Adult and pediatric participants were administered a single intravitreal (IVT) injection of rAAV2tYF-CB-hRS1, once in the study eye, at a dose of 3 x 10^11 vg/eye and followed for a minimum of 12 months after dose administration.
- rAAV2tYF-CB-hRS1 6 x 10^11 vg Per Eye: Group 3/4: Adult participants were administered a single intravitreal (IVT) injection of rAAV2tYF-CB-hRS1, once in the study eye, at a dose of 6 x 10^11 vg/eye and followed for a minimum of 12 months after dose administration.
Period: Overall Study
Arm/Group | rAAV2tYF-CB-hRS1 1 x 10^11 vg Per Eye | rAAV2tYF-CB-hRS1 3 x 10^11 vg Per Eye | rAAV2tYF-CB-hRS1 6 x 10^11 vg Per Eye
Started | 6 | 8 | 13
Completed Month 12 | 6 | 8 | 13
Started Long-Term Follow-Up | 6 | 8 | 13
Completed | 0 | 0 | 0
Not Completed | 6 | 8 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rAAV2tYF-CB-hRS1 1 x 10^11 vg Per Eye | rAAV2tYF-CB-hRS1 3 x 10^11 vg Per Eye | rAAV2tYF-CB-hRS1 6 x 10^11 vg Per Eye | Total
Number analyzed (Participants) | 6 | 8 | 13 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 5 | 0 | 6
  Between 18 and 65 years | 3 | 3 | 13 | 19
  >=65 years | 2 | 0 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 6 | 8 | 13 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 1 | 4
  Not Hispanic or Latino | 6 | 5 | 12 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 7 | 12 | 24
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Adverse Events
Description: Number of participants with ocular adverse events, assessed by standard ophthalmic examination, including slit lamp biomicroscopy, tonometry, and indirect ophthalmoscopy.
Time Frame: From Day 0 to Month 12 (12 months)
Population: All treated study participants with ocular treatment-emergent adverse events (TEAEs).
Measure: Count of Participants; unit: Participants
Arm/Group | rAAV2tYF-CB-hRS1 1 x 10^11 vg Per Eye | rAAV2tYF-CB-hRS1 3 x 10^11 vg Per Eye | rAAV2tYF-CB-hRS1 6 x 10^11 vg Per Eye
Number analyzed (Participants) | 6 | 8 | 13
Participants | 6 | 7 | 12

2. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA)
Description: Change in ETDRS (Early Treatment of Diabetic Retinopathy) Letter Score. Minimum value=0; Maximum value=100. Higher scores indicate better visual acuity. Change = 12 Mo value - Baseline value
Time Frame: From Day 0 to Month 12 (12 Months)
Population: All treated study participants with available data.
Measure: Mean (Standard Deviation); unit: ETDRS Letter Score
Arm/Group | rAAV2tYF-CB-hRS1 1 x 10^11 vg Per Eye | rAAV2tYF-CB-hRS1 3 x 10^11 vg Per Eye | rAAV2tYF-CB-hRS1 6 x 10^11 vg Per Eye
Number analyzed (Participants) | 6 | 8 | 12
ETDRS Letter Score
  Baseline Letter Score (Study Eye) | 38.7 (16.82) | 56.3 (8.65) | 50.4 (18.93)
  Month 12 Letter Score (Study Eye) | 39.5 (16.65) | 59.9 (10.29) | 51.4 (18.28)

3. Secondary Outcome: Change From Baseline in Schisis Cavity Size on Optical Coherence Tomography (OCT)
Description: Change in cystic cavity volume (mm^3), obtained from spectral domain optical coherence tomography (SD-OCT) of the retina, yielding volumetric measures of schisis cavity size and total cyst cavity. Change = 12 Mo value - Baseline value
Time Frame: From Day 0 to Month 12 (12 months)
Population: All treated study participants with available data.
Measure: Mean (Standard Deviation); unit: Cystic Cavity Volume (mm^3)
Arm/Group | rAAV2tYF-CB-hRS1 1 x 10^11 vg Per Eye | rAAV2tYF-CB-hRS1 3 x 10^11 vg Per Eye | rAAV2tYF-CB-hRS1 6 x 10^11 vg Per Eye
Number analyzed (Participants) | 6 | 7 | 10
Cystic Cavity Volume (mm^3)
  Baseline Cystic Cavity Volume (mm^3) (Study Eye) | 1.13 (1.34) | 1.12 (0.68) | 1.28 (1.57)
  Month12 Cystic Cavity Volume (mm^3) (Study Eye) | 1.33 (1.82) | 1.28 (0.62) | 1.04 (1.64)

4. Secondary Outcome: Change From Baseline in B-wave Amplitude in Electroretinogram (ERG) Responses
Description: Change in dark-adapted 3.0 B-wave amplitude (μV). Change = 12 Mo value - Baseline value
Time Frame: From Day 0 to Month 12 (12 months)
Population: All treated study participants with available data.
Measure: Mean (Standard Deviation); unit: μV
Arm/Group | rAAV2tYF-CB-hRS1 1 x 10^11 vg Per Eye | rAAV2tYF-CB-hRS1 3 x 10^11 vg Per Eye | rAAV2tYF-CB-hRS1 6 x 10^11 vg Per Eye
Number analyzed (Participants) | 6 | 6 | 10
μV
  Baseline Dark Adapted 3.0 B-Wave Amplitude (μV) | 107.3 (50.09) | 206.0 (60.95) | 169.9 (62.82)
  M12 Dark Adapted 3.0 B-Wave Amplitude (μV) | 92.8 (61.94) | 142.2 (62.77) | 164.0 (53.11)

ADVERSE EVENTS:
Time Frame: Study Day 0 through Month 12- Adverse Events; Study ongoing: adverse events beyond Month 12 to be updated at a later date
Arm/Group | rAAV2tYF-CB-hRS1 1 x 10^11 vg Per Eye | rAAV2tYF-CB-hRS1 3 x 10^11 vg Per Eye | rAAV2tYF-CB-hRS1 6 x 10^11 vg Per Eye
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8 | 0/13
Serious Adverse Events (participants affected / at risk) | 2/6 | 1/8 | 1/13
Other Adverse Events (participants affected / at risk) | 6/6 | 7/8 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rAAV2tYF-CB-hRS1 1 x 10^11 vg Per Eye (N=6) | rAAV2tYF-CB-hRS1 3 x 10^11 vg Per Eye (N=8) | rAAV2tYF-CB-hRS1 6 x 10^11 vg Per Eye (N=13)
Retinal detachment (Eye disorders) | 0 | 1 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0
Cerebellar stroke (Nervous system disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | rAAV2tYF-CB-hRS1 1 x 10^11 vg Per Eye (N=6) | rAAV2tYF-CB-hRS1 3 x 10^11 vg Per Eye (N=8) | rAAV2tYF-CB-hRS1 6 x 10^11 vg Per Eye (N=13)
Keratic precipitates (Eye disorders) | 2 | 2 | 7 — Ocular
Vitritis (Eye disorders) | 3 | 3 | 5 — Ocular
Anterior chamber cells (Eye disorders) | 0 | 2 | 8 — Ocular
Vitreous floaters (Eye disorders) | 0 | 2 | 6 — Ocular
Eye pain (Eye disorders) | 1 | 2 | 4 — Ocular
Vitreal cells (Eye disorders) | 1 | 1 | 5 — Ocular
Conjunctival haemorrhage (Eye disorders) | 2 | 2 | 3 — Ocular
Cataract subcapsular (Eye disorders) | 0 | 1 | 3 — Ocular
Vision blurred (Eye disorders) | 0 | 1 | 4 — Ocular
Vitreous haze (Eye disorders) | 0 | 1 | 4 — Ocular
Visual impairment (Eye disorders) | 0 | 2 | 2 — Ocular
Anterior chamber inflammation (Eye disorders) | 2 | 0 | 2 — Ocular
Retinal tear (Eye disorders) | 0 | 1 | 2 — Ocular
Anterior chamber flare (Eye disorders) | 0 | 1 | 2 — Ocular
Cataract (Eye disorders) | 0 | 0 | 3 — Ocular
Conjunctival hyperaemia (Eye disorders) | 1 | 0 | 2 — Ocular
Eye pruritus (Eye disorders) | 0 | 0 | 3 — Ocular
Photophobia (Eye disorders) | 0 | 1 | 2 — Ocular
Photopsia (Eye disorders) | 0 | 0 | 3 — Ocular
Lenticular opacities (Eye disorders) | 0 | 1 | 1 — Ocular
Conjunctival oedema (Eye disorders) | 0 | 2 | 0 — Ocular
Eyelid ptosis (Eye disorders) | 1 | 1 | 0 — Ocular
Iridocyclitis (Eye disorders) | 0 | 0 | 2 — Ocular
Lacrimation increased (Eye disorders) | 0 | 1 | 1 — Ocular
Ocular discomfort (Eye disorders) | 0 | 0 | 2 — Ocular
Retinal detachment (Eye disorders) | 0 | 1 | 1 — Ocular
Retinal haemorrhage (Eye disorders) | 0 | 1 | 1 — Ocular
Injection site haemorrhage (General disorders) | 1 | 2 | 3 — Ocular
Injection site discomfort (General disorders) | 0 | 1 | 1 — Ocular
Intraocular pressure (Investigations) | 1 | 1 | 2 — Ocular
Optic neuritis (Nervous system disorders) | 0 | 0 | 2 — Ocular
Pyrexia (General disorders) | 0 | 1 | 2 — Non-ocular
Feeling hot (General disorders) | 0 | 0 | 2 — Non-ocular
Blood pressure increased (Investigations) | 0 | 1 | 1 — Non-ocular
Weight increased (Investigations) | 0 | 0 | 2 — Non-ocular
White blood cell count increased (Investigations) | 0 | 1 | 1 — Non-ocular
Headache (Nervous system disorders) | 1 | 1 | 3 — Non-ocular
Viral upper respiratory tract infection (Infections and infestations) | 1 | 3 | 4 — Non-ocular
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 3 — Non-ocular
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 2 — Non-ocular
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 — Non-ocular
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 — Non-ocular
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 1 — Non-ocular
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 4 — Non-ocular
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 — Non-ocular
Increased appetite (Metabolism and nutrition disorders) | 1 | 0 | 3 — Non-ocular
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 — Non-ocular
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 — Non-ocular
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 — Non-ocular
Insomnia (Psychiatric disorders) | 0 | 1 | 3 — Non-ocular

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/22/NCT02416622/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-08): https://cdn.clinicaltrials.gov/large-docs/22/NCT02416622/SAP_001.pdf